CLINICAL TRIAL: NCT03571464
Title: Can Brief, Daily Training Using a Mobile Applications Help Change Maladaptive Beliefs? A Cross-over Randomized-control Study Evaluating the Efficacy of GGRO in Reducing Maladaptive Beliefs and Obsessive-compulsive Symptoms
Brief Title: Study of the Efficacy of GGRO: a Novel Cognitive Training App
Acronym: GGRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, María Roncero, Professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 706208
Record Dates: First submitted 2018-06-12; First posted 2018-06-27 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Obsessive Thoughts
Keywords: obsessive compulsive disorder; cognitive therapy; maladaptive beliefs; mobile app
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: All participants were requested to complete web-based assessment, with questionnaires relating to maladaptive beliefs, mood and OC symptoms at baseline (T1), 15 days following baseline (T2) and 30 days following baseline (T3). Participants in Immediate use GGRO group started using the app at baseline and continued using the app for 15 consecutive days. They were then requested to stop using the app until T3. Participants in the Delayed use GGRO group were requested to wait for 15 days and only then start using the app (cross-over) for 15 consecutive days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate use GGRO Mobile App (Experimental): The group starts using the GGRO Mobile App immediately after the first assessment (T1) for 15 days.
  Interventions: Device: GGRO Mobile App
- Delayed use GGRO Mobile App (Active Comparator): Delayed use GGRO Mobile App group started using the App 15 days after the first assessment (T2).
  Interventions: Device: GGRO Mobile App

INTERVENTIONS:
Device: GGRO Mobile App — GGRO was designed to challenge maladaptive beliefs that underlie common OCD symptoms (e.g., contamination, repugnant thoughts) as well as relationships obsessions. Users are presented with 'blocks' featuring statements such as "I take things as they come" or "Everything can end in a catastrophe". Users then have to respond to these statements by either pulling 'blocks' towards themselves (i.e., downwards) or throwing the blocks away from themselves (i.e., rejecting them upwards).

SUMMARY:
The aim of the present study was to evaluate the efficacy of GGRO reducing OCD related maladaptive beliefs and OCD symptoms. Specifically, a randomized controlled trial with crossover design was carried out in non-clinical population to assess pre-post changes in levels of OCD-related maladaptive beliefs and OCD symptoms, including relationship OCD (ROCD) symptoms, self-esteem, and depressive symptoms following 15 days of using GGRO.

DETAILED DESCRIPTION:
The implementation of Information and Communication Technologies in the treatment or prevention of OCD symptoms has been significantly lower compared to with its application in other anxiety disorders.

Recently, an exploratory study evaluated a brief, game-like, training exercise for challenging OCD-beliefs delivered via a mobile application platform named GGRO. However, more studies are needed to test the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Being a Spanish at native level, and having a mobile device capable of installing the application GGRO

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-09-25 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Change in obsessive beliefs | 15 days
  Score change in obsessive compulsive maladaptive beliefs measured by the short form of the Obsessive Beliefs Questionnaire (OBQ-20). Total score is computed as a mean of the 20 items, ranging from 1 "disagree very much" to 7 "agree very much". Higher scores indicate the person has more obsessive beliefs.

SECONDARY OUTCOMES:
Change in obsessive compulsive symptoms | 15 days
  Score change in obsessive-compulsive symptoms measured by the Obsessive Compulsive Inventory- Revised version (OCI-R). Total score is computed as a mean of the 18 items, ranging from 0 "not at all" to 4 "Extremely". Higher scores indicate a greater presence of obsessive-compulsive symptoms.
Change in depression symptoms | 15 days
  Score change in depression symptoms measured by Depression, Anxiety and Stres Scale (DASS). The depression scale is composed by the mean of 7 items, ranging from 0 "did not apply to me at all" to 3 "applied to me very much, or most of the time". Higher scores indicate a greater presence of obsessive -compulsive symptoms.
Change in Self-Esteem | 15 days
  Change in score of Single Ítem Self Esteem Scale (SISE). Self-Esteem is measured with this single item ranging from 1 "not very true for me" to 9 "very true for me". Higher scores indicates a higher Self-Esteem.

CONTACTS AND LOCATIONS:
Overall Officials: María Roncero, PhD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roncero M, Belloch A, Doron G. A novel approach to challenging OCD related beliefs using a mobile-app: An exploratory study. J Behav Ther Exp Psychiatry. 2018 Jun;59:157-160. doi: 10.1016/j.jbtep.2018.01.008. Epub 2018 Feb 2. PMID 29425951
- [Derived] Roncero M, Belloch A, Doron G. Can Brief, Daily Training Using a Mobile App Help Change Maladaptive Beliefs? Crossover Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Feb 13;7(2):e11443. doi: 10.2196/11443. PMID 30758294
- See also: Information about GGRO Mobile App and links to download — http://ggapps.net/2018/04/11/ggro-relationship-obsession-rocd/